CLINICAL TRIAL: NCT00031122
Title: The Spina Bifida Research Resource
Brief Title: Study of Genetic Risk Factors for Spina Bifida and Anencephaly
Acronym: SBRR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Laura. E. Mitchell, Ph.D., Institute for Biosciences and Technology, Texas A&M University
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 1R01HD039195-01 (NIH); 1R01HD039081-01 (NIH)
Record Dates: First submitted 2002-02-26; First posted 2002-02-27 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2009-05

CONDITIONS: Spina Bifida; Anencephaly
Keywords: Genetic Predisposition to Disease; Environmental Exposure; Chromosome Mapping; Data Collection
MeSH Terms: conditions — Spinal Dysraphism; Anencephaly; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA extracted from whole blood, saliva, buccal swab, and/or amniocytes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SBRR: Families with a child/pregnancy affected with spina bifida or anencephaly
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — There is no intervention in this study

SUMMARY:
The purpose of this study is to describe the genetic contribution to the neural tube defects spina bifida (SB) and anencephaly (A), which includes identifying patients, defining the roles of certain genes, and studying gene-environment interactions.

DETAILED DESCRIPTION:
The terms spina bifida and anencephaly include a range of developmental malformations that result from abnormal or incomplete closure of the neural tube. Despite advances in treatment and prenatal detection, these conditions remain as one of the most common and serious groups of birth defects. Spina bifida is associated with both increased mortality and morbidity, and anencephaly is always fatal. The occurrence of these conditions has a profound influence on affected individuals and their families and important public health implications. The etiology of NTDs has been of considerable interest for several decades. They are known to be etiologically heterogeneous and to occur in association with chromosome abnormalities, teratogenic exposures, and occasionally as part of single gene disorders. However, a specific causative agent cannot be identified in the vast majority of affected individuals. The etiology of NTDs in these "non-syndromic" patients is believed to be complex and to involve both genetic and environmental risk factors. Using a comprehensive research program, this study will evaluate the potential genetic determinants of SB and anencephaly in a large, well-characterized sample.

The family constellation used in this study consists of the proband (individual with an NTD - SB or A) and the proband's biologic parents and maternal grandparents. Blood or saliva samples are obtained from individuals and their families. Genomic DNA from all study participants is prepared from the samples, and genetic loci are evaluated. The proband, or his/her parents, complete a study questionnaire to obtain family history and epidemiologic information.

ELIGIBILITY:
Inclusion Criteria:

* Families that include at least 1 member who has SB or who had a fetus affected with SB or anencephaly

Exclusion Criteria:

* Have an NTD (SB or anencephaly) as a component of an identified syndrome
* Families of individuals who have diagnoses other than SB or anencephaly

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Volunteer participants recruited through support groups, clinics, and Web site responses
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2000-09; Primary Completion 2011-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Genetic loci identification and comparisons | After DNA sampling

CONTACTS AND LOCATIONS:
Overall Officials: Laura E. Mitchell, Ph.D., Principal Investigator — The Texas A & M University Health Science Center
Locations (2):
- United States (2):
  - The University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - The Texas A & M University Health Science Center, Houston, Texas